CLINICAL TRIAL: NCT03207204
Title: Long-term Clinical Evaluation of In-office Dental Bleaching Using a Violet Light (405-410 nm)
Brief Title: In-office Bleaching Using a Violet Light
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Patricia Moreira de Freitas, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 010
Record Dates: First submitted 2017-06-22; First posted 2017-07-02 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Tooth Bleaching; Dentin Sensitivity
Keywords: Dental bleaching; Color; Sensitivity; violet LED; Quality of life
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- G1 - 35% Hydrogen peroxide bleaching (Active Comparator): In-office bleaching performed with 35% hydrogen peroxide (4 sessions, 1 session/week);
  Interventions: Procedure: 35% Hydrogen peroxide bleaching
- G2 - 30% Carbamide peroxide bleaching (Active Comparator): In-office bleaching performed with 30% carbamide peroxide (4 sessions, 1 session/week);
  Interventions: Procedure: 30% Carbamide peroxide bleaching
- G3 - Violet LED bleaching 1 (Experimental): In-office bleaching performed with Violet LED (405-410 nm, 4 sessions, 1 session/week);
  Interventions: Procedure: Violet LED bleaching 1
- G4 - Violet LED bleaching 2 (Experimental): In-office bleaching performed with Violet LED (405-410 nm, 4 sessions, 2 sessions/week);
  Interventions: Procedure: Violet LED bleaching 2
- G5 - Photochemical protocol 1 (Experimental): In-office bleaching performed Violet LED associated to 35% hydrogen peroxide (4 sessions, 1 session / week);
  Interventions: Procedure: Photochemical protocol 1
- G6 - Photochemical protocol 2 (Experimental): In-office bleaching performed Violet LED associated to 30% carbamide peroxide (4 sessions, 1 session / week)
  Interventions: Procedure: Photochemical protocol 2
- G7 - Hybrid technique 1 (Experimental): hybrid technique HP (Violet LED + application of 35% hydrogen peroxide + violet LED) (4 sessions, 1 session/week)
  Interventions: Procedure: Hybrid technique 1
- G8 - Hybrid technique 2 (Experimental): Hybrid technique CP HP (Violet LED + application of 30% carbamide peroxide + violet LED) (4 sessions, 1 session/week).
  Interventions: Procedure: Hybrid technique 2

INTERVENTIONS:
Procedure: 35% Hydrogen peroxide bleaching — Application of 35% hydrogen peroxide on buccal face of anterior teeth (15-25). The application will be performed according to the manufacturer's instructions.
  Arms: G1 - 35% Hydrogen peroxide bleaching
Procedure: 30% Carbamide peroxide bleaching — Protocol: Application of 35% Carbamide peroxide on buccal face of anterior teeth (15-25). The application will be performed according to the manufacturer's instructions.
  Arms: G2 - 30% Carbamide peroxide bleaching
Procedure: Violet LED bleaching 1 — Protocol: Application of the Violet LED on buccal face of anterior teeth (15-25) with a distance of 8mm between the light source and teeth surface. The application will be performed for 60s, and then turned off for 30s. It will be repeated for 20x. The procedure will be performed 1 time a week.
  Arms: G3 - Violet LED bleaching 1
Procedure: Violet LED bleaching 2 — Protocol: Application of the Violet LED on buccal face of anterior teeth (15-25) with a distance of 8mm between the light source and teeth surface. The application will be performed for 60s, and then turned off for 30s. It will be repeated for 20x. The procedure will be performed 2 times a week.
  Arms: G4 - Violet LED bleaching 2
Procedure: Photochemical protocol 1 — Protocol: Application of 35% hydrogen peroxide on buccal face of anterior teeth (15-25). The application will be performed according to the manufacturer's instructions and associated with the application of Violet LED with a distance of 8mm between the light source and teeth surface. The application of Violet LED will be performed for 60s, and then turned off for 30s. It will be repeated for 20x. The procedure will be performed 1 time a week.
  Arms: G5 - Photochemical protocol 1
Procedure: Photochemical protocol 2 — Protocol: Application of 30% Carbamide peroxide on buccal face of anterior teeth (15-25). The application will be performed according to the manufacturer's instructions and associated with the application of Violet LED with a distance of 8mm between the light source and teeth surface. The application of Violet LED will be performed for 60s, and then turned off for 30s. It will be repeated for 20x. The procedure will be performed 1 time a week.
  Arms: G6 - Photochemical protocol 2
Procedure: Hybrid technique 1 — Protocol: Application of the Violet LED on buccal face of anterior teeth (15-25) with a distance of 8mm between the light source and teeth surface. The application will be performed for 60s, and then turned off for 30s. It will be repeated for 20x. In the last 10 illuminations of Violet LED it will be applied the 35% Hydrogen peroxide to act concomitantly with the light.
  Arms: G7 - Hybrid technique 1
Procedure: Hybrid technique 2 — Protocol: Application of the Violet LED on buccal face of anterior teeth (15-25) with a distance of 8mm between the light source and teeth surface. The application will be performed for 60s, and then turned off for 30s. It will be repeated for 20x. In the last 10 illuminations of Violet LED it will be applied the 30% Carbamide peroxide to act concomitantly with the light.
  Arms: G8 - Hybrid technique 2

SUMMARY:
The objective of this clinical study is to evaluate the effect of the whitening treatment performed with the violet LED light (405-410 nm), with or without a bleaching gel, on the tooth color changes (immediate and long-term), tooth sensitivity, satisfaction of participants in relation to the technique and impact on their quality of life. After being informed of the objectives of the study, 200 participants will be selected and randomly divided into a treatment group (n = 25): G1 - 35% hydrogen peroxide (HP) (4 sessions, 1 session/week); G2 - 30% carbamide peroxide (CP) (4 sessions, 1 session/week); G3 - Violet LED (405-410 nm, 4 sessions, 1 session/week); G4 - Violet LED (405-410 nm, 4 sessions, 2 sessions/week); G5 - Violet LED associated to 35% hydrogen peroxide (4 sessions, 1 session / week); G6 - Violet LED associated to 30% carbamide peroxide (4 sessions, 1 session / week); G7 - hybrid technique HP (Violet LED + application of 35% hydrogen peroxide + violet LED) (4 sessions, 1 session/week); G8 - Hybrid technique CP HP (Violet LED + application of 30% carbamide peroxide + violet LED) (4 sessions, 1 session/week). The color evaluation will be performed at predetermined times (before and immediately after treatment, 14 days after completion of bleaching and 3, 6 and 12 months after completion of bleaching), and quantitatively evaluated by colorimetric tests (objective and subjective) and spectrophotometry. In addition, it will be evaluated the tooth sensitivity during and after (48 hours) tooth whitening (VAS Scale), satisfaction with the treatment and impact on quality of life (OHIP-14 questionnaire). The data, except for survey data of satisfaction (descriptive evaluation), will be subjected to statistical analysis to determine the homogeneity and normality of the sample and for comparison between treatment groups, considering a 5% significance level.

DETAILED DESCRIPTION:
The objective of this clinical study is to evaluate the effect of the whitening treatment performed with the violet LED light (405-410 nm), with or without a bleaching gel, on the tooth color changes (immediate and long-term), tooth sensitivity, satisfaction of participants in relation to the technique and impact on their quality of life.

This study was approved by the research ethics committee of School of Dentistry of University of Sao Paulo (Protocol# 1.981.756). The experimental design is in according to CONSORT. The present research will be a blind, parallel and randomized study with similar allocation between the treatment groups. It will be included 200 participants, selected among the patients of the Special Laboratory of lasers in dentistry (LELO-FOUSP). After being being informed of the objectives of the study the participants will be randomly divided into a treatment group (n = 25):

G1 - In-office bleaching performed with 35% hydrogen peroxide (4 sessions, 1 session/week).

G2 - In-office bleaching performed with 30% carbamide peroxide (4 sessions, 1 session/week).

G3 - In-office bleaching performed with Violet LED (405-410 nm, 4 sessions, 1 session/week).

G4 - In-office bleaching performed with Violet LED (405-410 nm, 4 sessions, 2 sessions/week).

G5 - In-office bleaching performed Violet LED associated to 35% hydrogen peroxide (4 sessions, 1 session / week).

G6 - In-office bleaching performed Violet LED associated to 30% carbamide peroxide (4 sessions, 1 session / week).

G7 - hybrid technique HP (Violet LED + application of 35% hydrogen peroxide + violet LED) (4 sessions, 1 session/week).

G8 - Hybrid technique CP HP (Violet LED + application of 30% carbamide peroxide + violet LED) (4 sessions, 1 session/week).

The primary outcome of this study is the color alteration, which will be evaluated quantitatively by colorimetric (subjective) and spectrophotometric (objective) tests. Additionally, will be evaluated dental sensitivity during and after treatment (predetermined times), patient satisfaction regarding the treatment, and impact on patient quality of life (questionnaire OHIP-14).

The color measurement will be blind, in predetermined times (before the treatment, immediately after the treatment, 14 days after, 3 months after, 6 months after and 12 months after). It will be performed by two methods: subjectively, with a color scale; and objectively, with a clinical spectrophotometer.

The evaluation of dental sensitivity will be measured with a Visual analogue scale (VAS). It will be performed immediately after the treatment and 48 hours after the treatment.

The patient satisfaction regarding the treatment will be measured with a questionnaire for self-evaluation of the treatment, and will be applied 14 days after the end of treatment, 3 months after, 6 months after and 12 months after.

The evaluation of quality of life of the patients will be performed with the OHIP-14 questionnaire, which will be applied after the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of all the teeth, without restorations or caries on anterior teeth.
* Patients presenting the canine tooth color A3 (according to Vita classical scale) or darker.

Exclusion Criteria:

* Patients presenting systemic pathologies
* Patients presenting periodontal diseases
* Smokers or patients with systematic use of alcohol
* Patients presenting teeth with color alterations by tetracycline, fluorosis, endodontic treatments.
* Patients with historic of self-referenced sensitivity
* Pregnant or Breastfeeding period patients
* Presence of restorations on anterior teeth
* Patients presenting bruxism or systematic use of analgesics or anti-inflammatory drugs

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2017-07-02 (Actual); Primary Completion 2017-12-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Color alteration | 12 months after the treatment
  The color measurement will be blind, in predetermined time (12 months after the treatment). It will be performed with a clinical spectrophotometer.

SECONDARY OUTCOMES:
Dental sensitivity | Immediately after the treatment and 48 hours after the treatment
  The evaluation of dental sensitivity will be measured with a Visual analogue scale (VAS). It will be performed immediately after the treatment and 48 hours after the treatment.
Patient satisfaction regarding the treatment | 14 days after the end of treatment, 3 months after, 6 months after and 12 months after
  The patient satisfaction regarding the treatment will be measured with a questionnaire for self-evaluation of the treatment, and will be applied 14 days after the end of treatment, 3 months after, 6 months after and 12 months after.
Quality of life of the patients | Immediately after the end of bleaching
  The evaluation of quality of life of the patients will be performed with the OHIP-14 questionnaire, which will be applied after the end of the treatment.
Color change throughout 12 months with a visual color scale | Before, immediately after, 14 days, 3 months, 6 months and 12 months after bleaching
  The evaluation will be performed with a visual color scale
Color change throughout 6 months with a clinical spectrophotometer | Before, immediately after, 14 days, 3 months and 6 months after bleaching
  The evaluation will be performed with a clinical spectrophotometer

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Freitas, PhD, Study Chair — Associate Professor
Locations (1):
- School of Dentistry of USP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernardon JK, Sartori N, Ballarin A, Perdigao J, Lopes GC, Baratieri LN. Clinical performance of vital bleaching techniques. Oper Dent. 2010 Jan-Feb;35(1):3-10. doi: 10.2341/09-008CR. PMID 20166405
- [Background] Boushell LW, Ritter AV, Garland GE, Tiwana KK, Smith LR, Broome A, Leonard RH. Nightguard vital bleaching: side effects and patient satisfaction 10 to 17 years post-treatment. J Esthet Restor Dent. 2012 Jun;24(3):211-9. doi: 10.1111/j.1708-8240.2011.00479.x. Epub 2011 Oct 11. PMID 22691084